

CorEvitas Statistical Analysis Plan: Analysis of tofacitinib initiators with PsA:

Phase II Follow-up Analysis

Prepared for: Pfizer

Prepared by: PPD , MS

9 December 2021

### Title: Analysis of tofacitinib initiators with PsA

Overall Aim: To describe baseline demographic, therapy history, and disease activity characteristics and assess change in disease activity measures six months after initiation of tofacitinib

To accomplish the overall aim, we will:

- Objective 1: Summarize patient characteristics at baseline and calculate changes in various disease activity measures over time among all eligible initiators of tofacitinib
- Objective 2: Summarize patient characteristics at baseline and calculate changes in various disease activity measures separately for monotherapy and combination therapy initiators, and compare these groups

#### Definitions:

- Oral small molecules (OSMs): methotrexate, leflunomide, sulfasalazine, apremilast
- Tofacitinib monotherapy: initiation of tofacitinib with no other (pre-existing or new) DMARD prescriptions
- Tofacitinib combination therapy: initiation of tofacitinib with a concomitant (pre-existing or new) prescription of at least one OSM

# Registry description:

CorEvitas' Psoriatic Arthritis/Spondyloarthropathy Registry is a prospective, multicenter, observational disease—based registry that was started March 2013.

From initiation until April 2017, inclusion criteria in the registry were as follows:

- Meet diagnostic criteria for psoriatic arthritis (PsA), ankylosing spondylitis (AS), axial or peripheral SpA
- Age ≥ 18 years of age as of the patient's PsA/SpA diagnosis
- Subject must be able and willing to provide consent

From April 2017 until February 2018, the inclusion criteria were modified as follows:

- Meet diagnostic criteria for ankylosing spondylitis (AS), axial or peripheral SpA or PsA
- Age ≥ 18 years of age as of the patient's PsA/SpA diagnosis
- Subjects needed to be diagnosed with psoriatic arthritis (PsA) by their rheumatologist or meet the modified New York classification criteria for ankylosing spondylitis (AS)
- Subjects needed to be a newly prescribed (first time) user of an FDA-approved eligible biologic for the treatment of PsA or AS at time of enrollment. Eligible biologics for inclusion in the registry include abatacept, adalimumab, certolizumab, etanercept, golimumab, infliximab, secukinumab, ustekinumab (only FDA approved for PsA).

From February 2018 until October 2018, the inclusion criteria were modified as follows:

- Non-biologic medications have been added as eligible medications for enrollment of patients diagnosed with Psoriatic Arthritis.
- Eligibility for Psoriatic Arthritis patients has been expanded to include patients currently on an eligible medication at the time of enrollment.

From October 2018 until August 2019, the enrollment criteria were modified as follows:

- For PsA patients, only incident users (either prescribed or actually receiving first dose on the day
  of the enrollment visit) of eligible medications are eligible. Patients who are prevalent users
  (currently receiving a medication or first dose received prior to the enrollment visit) are no
  longer eligible for new enrollment.
- 1:2 enrollment ratio is defined as one (1) IL-17 inhibitor or JAK-inhibitor to every two (2) biologics.

From August 2019 forward, the enrollment criteria were expanded as follows:

- Apremilast (Otezla) has been added as an eligible medication at enrollment.
- Eligible diagnoses at enrollment will now include PsA, AS (per modNY), or Axial Spondyloarthritis (per ASAS), radiographic or non-radiographic.

CorEvitas patients and their rheumatologists complete questionnaires, including information on laboratory measurements and radiographic results from routine visits, at approximately 6-month intervals.

# Study Cohort:

For this analysis, the eligible population will be selected using the following criteria:

- Have a diagnosis of PsA
- Initiate tofacitinib monotherapy or in combination with OSMs (pre-existing or concurrent) during or after December 2017
- Have a follow-up visit occurring six (± 3) months after initiation

Initiators will be ineligible for analysis if:

Any initiations result in a combination of tofacitinib with TNFi or non-TNFi bDMARDs, whether multiple initiations occur at the same time or a new therapy is added to an existing regimen

# Analysis:

# Milestone 1:

Consider the demographic, patient, and disease characteristics of all eligible tofacitinib initiators in **Table 1**. Categorical variables will be examined using frequencies and proportions. Continuous variables will be summarized using descriptive statistics (mean, standard deviation, minimum, 25% percentile, median, 75% percentile, maximum).

In Table 2, we will present the therapy status of initiators at the six-month follow-up visit.

**Table 3** will examine the outcomes of interest at the six-month follow-up visit. Binary outcomes will be presented as response rates with 95% CI using normal approximation to binomial proportions, and summary statistics (n, mean (SD), [P0,P25,P50,P75,P100]) baseline, six-month, and change in continuous outcomes will also be presented.

# Milestone 2:

The analyses stratified by mono- and combination therapy for this milestone will be completed when the sample reaches at least 100 initiators in both mono- and combination therapy groups.

Consider the demographic, patient, and disease characteristics of the tofacitinib monotherapy and combination therapy initiators in **Table 4**. Categorical variables will be examined using frequencies and proportions, and, when sample size allows for significance testing, differences across therapy patterns will be tested using chi-square or Fisher exact tests. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, minimum, 25% percentile, median, 75% percentile, maximum). When sample size allows for significance testing, differences across therapy groups will be tested using Wilcoxon rank sum tests.

In Table 5, we will present the therapy status of initiators at the six-month follow-up visit.

Table 6 will examine the outcomes of interest at the six-month follow-up visit. The change from baseline to six months in continuous outcomes will be analyzed using an analysis of covariance model with fixed effects for treatment group and baseline value. For continuous outcomes, we will not impute missing values. Also, for those discontinuing therapy prior to follow-up, we will use the value immediately prior to discontinuation as the follow-up value. We will present LS Means (standard error) for each therapy group as well as the difference in the LS Means (standard error), 95% CI and p-value. Binary outcomes will be presented as response rates with 95% CIs using normal approximation to binomial proportions. We will provide comparisons of response rates between groups with 95% CIs and p-values using normal approximation for the difference in binomial proportions. As a supportive analysis, treatment difference between the groups will be assessed using logistic regression models with treatment group as the sole covariate. For binary outcomes, we will impute non-response for missing values and for those patients discontinuing therapy prior to follow-up.

In **Table 7**, we will present summary statistics (n, mean (SD), [P0,P25,P50,P75,P100]) for continuous outcomes featured in Table 3 at baseline, six months, and the difference from baseline to six months overall and by therapy group.

#### Characteristics of Interest:

The following characteristics will be assessed on index date:

- Age
- Sex
- Race
- Work status
- BMI (continuous and categorical)
- Duration of PsA symptoms
- Time since PsA diagnosis
- Time since onset of PsO
- Physician-reported comorbidity history

- Cerebro-cardiovascular disease (CVD) <sup>a</sup>
- Depression
- Diabetes mellitus
- Any cancer (excluding NMSC)
- NMSC
- HTN
- Hyperlipidemia
- Crohn's disease
- Anxiety
- Psoriasis
- Fibromyalgia
- Serious infections b
- Metabolic syndrome
- Ulcerative colitis
- Uveitis
- Smoking status
  - Former, Current, Never
  - Number cigarettes smoked per day
  - Smoking duration
- Alcohol use
  - Yes/No
  - Number drinks per week
- Therapy history
  - History of prior biologic use
  - History of prior TNFi use
  - History of prior non-TNFi bDMARD use
  - History of prior OSM use
  - Current OSM use
    - Current MTX use
  - Current NSAID use
  - o Current opioid use
  - Current aspirin use
  - Current prednisone use
- Disease activity measures
  - Tender joint count (28 and 68)
  - Swollen joint count (28 and 66)
  - Enthesitis
  - SPARCC count
  - LEI count
  - Dactylitis
  - Dactylitis count
  - Nail VAS
  - o BSA (continuous and categorical)
  - o CRP
  - ESR
  - Clinical global assessment of PsO (continuous and categorical).
- Composite measures
  - MDA

- DAPSA (continuous and categorical)
- cDAPSA (continuous and categorical)
- PASDAS
- CDAI (continuous and categorical)
- Patient reported outcome measures
  - Patient pain
  - Patient-reported fatigue
  - Patient global skin assessment
  - HAQ-DI
  - HAQ-S
  - o EQ-5D
  - WPAI domains (4 categories)
- Psoriatic nail dystrophy
- Spinal mobility measures
  - Occiput to wall distance
  - Modified Schober

At the six-month follow-up visit, the following will be assessed:

Among those not in the specified disease activity state, achievement of:

- Minimal Disease Activity
- Body Surface Area Score of 0
- PASDAS < 3.2</li>
- Resolution of enthesitis
- Resolution of dactvlitis
- Clinical Global Assessment of PsO achievement of "Clear" or "Almost Clear"

# Baseline to six months change in:

- cDAPSA
- DAPSA
- PASDAS
- HAQ-DI
- Low Disease Activity as defined by cDAPSA (cDAPSA ≤ 13)
- BSA
- CDAI
- Tender joint count (68)
- Swollen joint count (66)
- Patient global skin assessment
- Patient pain
- Patient fatigue
- Clinical Global Assessment of PsO
- WPAI Domains

<sup>\*</sup> CVD includes: cardiac revascularization procedure (CABG, stent, angioplasty), ventricular arrhythmia, cardiac arrest, myocardial infarction, acute coronary syndrome, unstable angina, other coronary artery disease, CHF (with and without hospitalization), stroke, transient ischemic attack, other CV, deep vein thrombosis, peripheral arterial disease, pulmonary embolism, and carotid artery disease

<sup>&</sup>lt;sup>b</sup> Serious infections include: joint bursa infection, cellulitis, sinusitis, candida, diverticulitis, sepsis, pneumonia, bronchitis, gastroenteritis, meningitis, urinary tract infection, upper respiratory infection, tuberculosis, and other infection

# Feasibility Assessment and Projections:

Using the October 1, 2021 version of the PsA registry, we have identified the following therapy patterns among initiators of tofacitinib

| | Eligible Initiations, N (%) |
|-----------------------------|-----------------------------|
| All tofacitinib initiations | 213 |
| Monotherapy | 132 (62.0) |
| Combination with OSMs only | 81 (38.0) |
| Combination with MTX | 58 (71.6) |

| | Monotherapy Combination with OSMs | |
|---------------------|-----------------------------------|------------|
| Eligible Initiators | 132 | 81 |
| Six-month visit | 59 (44.7%) | 55 (67.9%) |

# **Shell Tables**

Table 1. Patient demographic characteristics among all tofacitinib initiators

| All Patients, N | Overall |
|---|---|
| Age (years), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Female, n/N (%) | |
| Race, n/N (%) | |
| White | |
| Black | |
| Asian | |
| Other | |
| Work Status, n/N (%) | |
| Full Time/Part Time | |
| Retired | |
| Disabled | |
| Other | |
| BMI (kg/m²), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| BMI Category (kg/m²), n/N (%) | |
| < 25 | |
| 25 to < 30 | |
| 30 + | |
| Duration of PsA Symptoms (years), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Time Since PsA Diagnosis (years), n, Mean (SD), [P0,P25,P50,P75,P100] | |

| All Patients, N | Overall |
|-------------------------------------------------------------------|---------|
| Time Since PsO Onset (years), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Psoriasis, n/N (%) | |
| Psoriatic Nail Dystrophy, n/N (%) | |
| History of Comorbidities, n/N (%) | |
| CVDb | |
| Depression | |
| Diabetes | |
| Malignancy <sup>c</sup> | |
| NMSC | |
| Hypertension | |
| Hyperlipidemia | |
| Crohns Disease | |
| Anxiety | |
| Fibromyalgia | |
| Serious Infections <sup>d</sup> | |
| Metabolic Syndrome | |
| Ulcerative Colitis | |
| Uveitis | |
| Smoking Status, n/N (%) | |
| Never | |
| Previous | |
| Current | |
| Cigarettes per day, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Smoking duration, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Alcohol Use, n/N (%) | |
| Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Number of Prior Biologics, n/N (%) | |
| 0 | |
| 1 | |
| 2+ | |
| Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Number of Prior TNFs, n/N (%) | |
| 0 | |
| 1 | |
| 2+ | |
| Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Number of Prior non-TNFs, n/N (%) | |

| All Patients, N | Overall |
|--------------------------------------------------------------|---------|
| 0 | |
| 1 | |
| 2+ | |
| Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Number of Prior OSMs, n/N (%) | |
| 0 | |
| 1 | |
| 2 + | |
| Current OSM Use, n/N (%) | |
| Current MTX Use, n/N (%) | |
| Current NSAID Use, n/N (%) | |
| Current Opioid Use, n/N (%) | |
| Current Aspirin Use, n/N (%) | |
| Prednisone Use, n/N (%) | |
| None | |
| Missing Dose | |
| Dose < 10 mg | |
| Dose ≥ 10 mg | |
| Tender Joints (28), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Tender Joints (68), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Swollen Joints (28), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Swollen Joints (66), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Enthesitis, n/N (%) | |
| SPARCC Enthesitis Count, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| LEI Count, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Dactylitis, n/N (%) | |
| Dactylitis Count, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| CDAI, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| CDAI Category, n/N (%) | |
| Remission (CDAI ≤ 2.8) | |
| Low (2.8 < CDAI ≤ 10) | |
| Moderate (10 < CDAI ≤ 22) | |
| High (22 < CDAI) | |
| Minimal Disease Activity, n/N (%) | |
| DAPSA, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| DAPSA Category, n/N (%) | |
| DAPSA ≤ 4 | |
| 4 < DAPSA ≤ 14 | |

| All Patients, N | Overall |
|---|---|
| 14 < DAPSA ≤ 28 | |
| 28 < DAPSA | |
| cDAPSA, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| cDAPSA Category, n/N (%) | |
| cDAPSA ≤ 3 | |
| 3 < cDAPSA ≤ 13 | |
| 13 < cDAPSA ≤ 27 | |
| 27 < cDAPSA | |
| PASDAS, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| PASDAS ≤ 3.2 | |
| 3.2 < PASDAS ≤ 4.2 | |
| 4.2 < PASDAS ≤ 6 | |
| 6 < PASDAS | |
| Nail VAS, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Body Surface Area (%), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| BSA Category (%), n/N (%) | |
| 0 | |
| > 0 to < 3 | |
| 3 to < 10 | |
| ≥ 10 | |
| CRP (mg/L), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| ESR (mm/hr), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Patient Pain (0-100 VAS), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Patient Fatigue (0-100 VAS), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Patient Global Skin Assessment (0-100 VAS), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Clinical Global Assessment of PsO <sup>1</sup> , n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Clinical Global Assessment of PsO <sup>1</sup> Category, n/N (%) | |
| Clear/Almost Clear | |
| Mild | |
| Moderate | |
| Severe | |
| HAQ-DI, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| HAQ-S, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| EQ-5D, n, Mean (SD), [P0,P25,P50,P75,P100] | |
| WPAI Domains (%), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Work Time Missed | |
| Impairment While Working | |
| Overall Work Impairment | |

| All Patients, N | Overall |
|--------------------------------------------------------------------|---------|
| Activity Impairment | |
| Spinal Mobility Measures (cm), n, Mean (SD), [P0,P25,P50,P75,P100] | |
| Occiput to Wall Distance | |
| Modified Schober | |

SD = standard deviation, P0 = minimum, P25 = 25th percentile, P50 = median, P75 = 75th percentile, P100 = maximum

Table 2. Therapy status six months post-initiation

| | Overall |
|----------------------------------------------|---------|
| All Patients, N | |
| Remain on tofacitinib, n (%) | |
| Discontinued tofacitinib, n (%) <sup>a</sup> | |
| Switched to a bDMARD, n (%) <sup>b</sup> | |

This group consists of those discontinuing tofacitinib and not initiating a bDMARD at or prior to the six-month follow-up visit

Table 3. Summary statistics of continuous outcomes at baseline, six months, and change from baseline to six months

| | Overall |
|---|---|
| All Initiators, N | |
| Achievement of: | Response Rate (95% CI) |
| LDA (cDAPSA) | |
| Minimal Disease Activity | |
| Body Surface Area Score of 0 | |
| PASDAS < 3.2 | |
| Resolution of enthesitis | |
| Resolution of dactylitis | |
| Clinical Global Assessment of PsO – Clear or Almost Clear | |

<sup>&</sup>lt;sup>a</sup> p-values from chi-square or Fisher exact tests for categorical variables and from Wilcoxon rank-sum tests for continuous variables, included for descriptive purposes only

<sup>&</sup>lt;sup>b</sup> History of cardiovascular disease includes history of: hypertension, hyperlipidemia, cardiac revascularization procedure (CABG, stent, angioplasty), ventricular arrythmia, cardiac arrest, myocardial infarction, acute coronary syndrome, unstable angina, CHF (with and without hospitalization), stroke, transient ischemic attack, other CV, deep vein thrombosis, peripheral arterial disease, peripheral arterial thrombosis, urgent peripheral revascularization, peripheral ischemia/gangrene, pulmonary embolism, carotid artery disease, and hemorrhage.

<sup>&</sup>lt;sup>c</sup> Malignancy includes breast cancer, lung cancer, lymphoma, skin cancer (squamous cell), and other cancers.

d Serious infections include the following: joint/bursa infection, cellulitis, sinusitis, diverticulitis, sepsis, pneumonia, bronchitis, gastroenteritis, meningitis, urinary tract infection, upper respiratory infection, tuberculosis, and other infections.

e Biologics: Humira, Enbrel, Cimzia, Simponi, Remicade, Orencia, Taltz, Cosentyx, Stelara

<sup>&</sup>lt;sup>1</sup> TNFs: Humira, Enbrel, Cimzia, Simponi, Remicade

non-TNFs: Orencia, Taltz, Cosentyx, Stelara

h cDMARDs: MTX, Arava, Azulfidine, Otezla

<sup>&</sup>lt;sup>1</sup> Clinical Global Assessment of PsO is scored on a five-point scale from 0-4, with corresponding interpretations of Clear, Almost Clear, Mild, Moderate, and Severe, respectively.

This group consists of those discontinuing tofacitinib and initiating a bDMARD at or prior to the six-month follow-up visit

| | Overall |
|--------------------------------|------------------------------------|
| | n, mean (SD), [P0,P25,P50,P75,P100 |
| cDAPSA | Baseline |
| | Six Months |
| | Difference a |
| DAPSA | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| PASDAS | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| HAQ-DI | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| BSA | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| CDAI | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Tender joint count (68) | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Swollen joint count (66) | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Patient global skin assessment | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Patient pain | Baseline |
| • | Six Months |
| | Difference <sup>a</sup> |
| Patient fatigue | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |

| | Overall |
|-----------------------------------|-------------------------|
| Clinical Global Assessment of PsO | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Work time missed | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Impairment while working | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Overall work impairment | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |
| Activity impairment | Baseline |
| | Six Months |
| | Difference <sup>a</sup> |

a Calculated as six-month value minus baseline value

**Table 4.** Patient demographic characteristics by monotherapy and combination therapy, among all tofacitinib initiators

| | Overall | Mono | Combo | p-value |
|---|---|---|---|---|
| All Patients, N | | | | |
| Age (years), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Female, n/N (%) | | | | |
| Race, n/N (%) | | | | |
| White | | | | |
| Black | | | | |
| Asian | | | | |
| Other | | | | |
| Work Status, n/N (%) | | | | |
| Full Time/Part Time | | | | |
| Retired | | | | |
| Disabled | | | | |
| Other | | | | |
| BMI (kg/m²), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| BMI Category (kg/m²), n/N (%) | | | | |
| < 25 | | | | |
| 25 to < 30 | | | | |
| 30 + | | | | |
| Duration of PsA Symptoms (years), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Time Since PsA Diagnosis (years), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Time Since PsO Onset (years), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Psoriasis, n/N (%) | | | | |
| Psoriatic Nail Dystrophy, n/N (%) | | | | |
| History of Comorbidities, n/N (%) | | | | |
| CVDp | | | | |
| Depression | | | | |
| Diabetes | | | | |
| Malignancy <sup>c</sup> | | | | |
| NMSC | | | | |
| Hypertension | | | | |
| Hyperlipidemia | | | | |
| Crohns Disease | | | | |
| Anxiety | | | | |
| Fibromyalgia | | | | |
| Serious Infections <sup>d</sup> | | | | |
| Metabolic Syndrome | | | | |

| Ulcerative Colltis Uveitis Smoking Status, n/N (%) Never Previous Current Cigarettes per day, n, Mean (SD), [P0,P25,P50,P75,P100] Smoking Duration, n, Mean (SD), [P0,P25,P50,P75,P100] Alcohol Use, n/N (%) Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2+ Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2+ Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2+ Prior SMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior ono-TNFs, n/N (%) 0 1 2+ Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2+ Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current NSAID Use, n/N (%) Current NSAID Use, n/N (%) Current NSAID Use, n/N (%) Prednisone Use, n/N (%) Prednisone Use, n/N (%) | verall Mono | Combo | p-value |
|---|---|---|---|
| Never | | | |
| Never | | | |
| Previous Current Cigarettes per day, n, Mean (SD), [P0,P25,P50,P75,P100] Smoking Duration, n, Mean (SD), [P0,P25,P50,P75,P100] Alcohol Use, n/N (%) Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Current Cigarettes per day, n, Mean (SD), [P0,P25,P50,P75,P100] Smoking Duration, n, Mean (SD), [P0,P25,P50,P75,P100] Alcohol Use, n/N (%) Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Osm Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Cigarettes per day, n, Mean (SD), [P0,P25,P50,P75,P100] Smoking Duration, n, Mean (SD), [P0,P25,P50,P75,P100] Alcohol Use, n/N (%) Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current NSAID Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Opioid Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Smoking Duration, n, Mean (SD), [P0,P25,P50,P75,P100] Alcohol Use, n/N (%) Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current MTX Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Alcohol Use, n/N (%) Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Number drinks per week, n, Mean (SD), [P0,P25,P50,P75,P100] Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Prior Biologics, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior Biologics, n/N (%) 0 1 2+ Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2+ Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2+ Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2+ Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2+ Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Number of Prior Biologics, n/N (%) 0 1 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 0 1 2+ Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2+ Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2+ Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2+ Current OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 Current MTX Use, n/N (%) Current MTX Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 1 2+ Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2+ Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2+ Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2+ Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2+ Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Current Aspirin Use, n/N (%) | | | |
| 2 + Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Prior TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior TNFs, n/N (%) 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Aspirin Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Number of Prior TNFs, n/N (%) 0 1 2+ Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2+ Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2+ Current OF Prior OSMs, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 0 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 1 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 2 + Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Prior non-TNFs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Number of Prior non-TNFs, n/N (%) 0 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 0 1 2+ Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2+ Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 1 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 2 + Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Prior OSMs, n, Mean (SD), [P0,P25,P50,P75,P100] Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Number of Prior OSMs, n/N (%) 0 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 0 1 2+ Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 1 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| 2 + Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Current OSM Use, n/N (%) Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Current MTX Use, n/N (%) Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Current NSAID Use, n/N (%) Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Current Opioid Use, n/N (%) Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Current Aspirin Use, n/N (%) Prednisone Use, n/N (%) | | | |
| Prednisone Use, n/N (%) | | | |
| None | | | |
| None | | | |
| Missing Dose | | | |

| | Overall | Mono | Combo | p-value |
|---|---|---|---|---|
| Dose < 10 mg | | | | |
| Dose ≥ 10 mg | | | | |
| Tender Joints (28), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Tender Joints (68), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Swollen Joints (28), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Swollen Joints (66), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Enthesitis, n/N (%) | | | | |
| SPARCC Enthesitis Count, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| LEI Count, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Dactylitis, n/N (%) | | | | |
| Dactylitis Count, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| CDAI, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| CDAI Category, n/N (%) | | | | |
| Remission (CDAI ≤ 2.8) | | | | |
| Low (2.8 < CDAI ≤ 10) | | | | |
| Moderate (10 < CDAI ≤ 22) | | | | |
| High (22 < CDAI) | | | | |
| Minimal Disease Activity, n/N (%) | | | | |
| DAPSA, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| DAPSA Category, n/N (%) | | | | |
| DAPSA ≤ 4 | | | | |
| 4 < DAPSA ≤ 14 | | | | |
| 14 < DAPSA ≤ 28 | | | | |
| 28 < DAPSA | | | | |
| cDAPSA, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| cDAPSA Category, n/N (%) | | | | |
| cDAPSA ≤ 3 | | | | |
| 3 < cDAPSA ≤ 13 | | | | |
| 13 < cDAPSA ≤ 27 | | | | |
| 27 < cDAPSA | | | | |
| PASDAS, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Nail VAS, n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| Body Surface Area (%), n, Mean (SD), [P0,P25,P50,P75,P100] | | | | |
| BSA Category (%), n/N (%) | | | | |
| 0 | | | | |
| > 0 to < 3 | | | | |
| 3 to < 10 | | | | |
| ≥ 10 | | | | |
| | | - | | |

| p-value |
|---------|

SD = standard deviation, P0 = minimum, P25 = 25th percentile, P50 = median, P75 = 75th percentile, P100 = maximum

<sup>&</sup>lt;sup>a</sup> p-values from chi-square or Fisher exact tests for categorical variables and from Wilcoxon rank-sum tests for continuous variables, included for descriptive purposes only

b History of cardiovascular disease includes history of: hypertension, hyperlipidemia, cardiac revascularization procedure (CABG, stent, angioplasty), ventricular arrythmia, cardiac arrest, myocardial infarction, acute coronary syndrome, unstable angina, CHF (with and without hospitalization), stroke, transient ischemic attack, other CV, deep vein thrombosis, peripheral arterial disease, peripheral arterial thrombosis, urgent peripheral revascularization, peripheral ischemia/gangrene, pulmonary embolism, carotid artery disease, and hemorrhage.

<sup>&</sup>lt;sup>c</sup> Malignancy includes breast cancer, lung cancer, lymphoma, skin cancer (squamous cell), and other cancers.

d Serious infections include the following: joint/bursa infection, cellulitis, sinusitis, diverticulitis, sepsis, pneumonia, bronchitis, gastroenteritis, meningitis, urinary tract infection, upper respiratory infection, tuberculosis, and other infections.

Biologics: Humira, Enbrel, Cimzia, Simponi, Remicade, Orencia, Taltz, Cosentyx, Stelara

<sup>&</sup>lt;sup>1</sup> TNFs: Humira, Enbrel, Cimzia, Simponi, Remicade

<sup>&</sup>lt;sup>9</sup> non-TNFs: Orencia, Taltz, Cosentyx, Stelara

h cDMARDs: MTX, Arava, Azulfidine, Otezla

<sup>&</sup>lt;sup>1</sup> Clinical Global Assessment of PsO is scored on a five-point scale from 0-4, with corresponding interpretations of Clear, Almost Clear, Mild, Moderate, and Severe, respectively.

Table 5. Therapy status six months post-initiation

| | Overall | Mono | Combo | p-value ª |
|---|---|---|---|---|
| All Patients, N | | | | |
| Remain on tofacitinib, n (%) | | | | |
| Discontinued tofacitinib, n (%) <sup>b</sup> | | | | |
| Switched to a bDMARD, n (%) ° | | | | |
| Added OSM, n (%) | | | | |
| Discontinued OSM, n (%) | | | | |

a p-value from chi-square test

<sup>&</sup>lt;sup>b</sup> This group consists of those discontinuing tofacitinib and not initiating a bDMARD at or prior to the six-month follow-up visit

<sup>&</sup>lt;sup>c</sup> This group consists of those discontinuing tofacitinib and initiating a bDMARD at or prior to the six-month follow-up visit

090177e199407874\Final\Final On: 02-Feb-2022 15:52 (GMT)

Table 6. Disease activity outcomes at six months

| | Mono | Combo | Mono vs Combo | | |
|---|---|---|---|---|---|
| Binary Outcomes | Response Rate<br>(95% CI) <sup>a</sup> | Response Rate<br>(95% CI) <sup>a</sup> | Rate Difference<br>(95% CI) <sup>a</sup> | p-value <sup>a</sup> | OR<br>(95% CI) |
| Achievement of: | | | | | |
| LDA (cDAPSA) | | | | | |
| Minimal Disease Activity | | | | | |
| Body Surface Area Score of 0 | | | | | |
| PASDAS < 3.2 | | | | | |
| Resolution of enthesitis | | | | | |
| Resolution of dactylitis | | | | | |
| Clinical Global Assessment of PsO –<br>Clear or Almost Clear | | | | | |
| Continuous Outcomes | LS Means (SE) | LS Means (SE) | Δ LS Means<br>(SE) 95% CI | | |
| Baseline to six-month change in: | | | | | |
| cDAPSA | | | | | |
| DAPSA | | | | | |
| PASDAS | | | | | |
| HAQ-DI | | | | | |
| BSA | | | | | |
| CDAI | | | | | |
| Tender joint count | | | | | |
| Swollen joint count | | | | | |
| Patient global skin assessment | | | | | |
| Patient pain | | | | | |
| Patient fatigue | | | | | |
| Clinical Global Assessment of PsO | | | | | |
| Work Time Missed | | | | | |
| Impairment While Working | | | | | |
| Overall Work Impairment | | | | | |
| Activity Impairment | | | | | |

<sup>&</sup>lt;sup>a</sup> 95% CI for the response rate and 95% CI and p-value for the rate difference were based on normal approximation to binomial proportions. OR (95% CI) was based on a logistic regression model with treatment group as the sole covariate

**Table 7.** Summary statistics of continuous outcomes at baseline, six months, and change from baseline to six months

| | | Overall | Mono | Combo |
|---|---|---|---|---|
| All Initiators, N | | | | |
| Continuous Outcome, n, mean (SD),<br>[P0,P25,P50,P75,P100] | | | | |
| cDAPSA | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| DAPSA | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| PASDAS | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| HAQ-DI | Baseline | | | |
| HAQ-DI BSA CDAI Tender joint count (68) | Six Months | | | |
| • | Difference <sup>a</sup> | | | |
| BSA | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| CDAI | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| Tender joint count (68) | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| Swollen joint count (66) | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| Patient global skin assessment | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| Swollen joint count (66) Patient global skin assessment Patient pain | Baseline | | | |
| | Six Months | | | |
| | Difference a | | | |

| | | Overall | Mono | Combo |
|---|---|---|---|---|
| Patient fatigue | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| Clinical Global Assessment of PsO | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| Work time missed | Baseline | | | |
| | Six Months | | | |
| | Difference a | | | |
| Impairment while working | Baseline | | | |
| | Six Months | | | |
| | Difference <sup>a</sup> | | | |
| Overall work impairment | Baseline | | | |
| | Six Months | | | |
| | Difference a | | | |
| Activity impairment | Baseline | | | |
| , i | Six Months | | | |
| Activity impairment | Difference <sup>a</sup> | | | |

a Calculated as six-month value minus baseline value